CLINICAL TRIAL: NCT00685542
Title: Phase IV Study of Diacerein in Human Hand Osteoarthritis
Brief Title: Effect of Diacerein on Hand Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Myungmoon Pharm. Co. (Unknown)
Responsible Party: Seoul National University Hopital, Eun Bong Lee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-081-043-232
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Osteoarthritis
Keywords: diacerein; osteoarthritis; hand
MeSH Terms: conditions — Osteoarthritis | interventions — diacerein; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Diacerein 50mg bid
  Interventions: Drug: diacerein
- 2 (Placebo Comparator): placebo 50mg bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: diacerein — Diacerein 50mg bid
  Other Names: Atrodar 50mg bid
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Ostearthritis is one of the most common arthritis, affecting more than 30% of aged people world-widely. The disease is characterized by pain and stiffness of the affected joints and is the most common cause of disability in aged people. It commonly affects knee, hip, hand and spine joints. Diacerein is a drug developed specifically for the treatment of osteoarthritis. It has inhibitory effects on interleukin-1 (IL-1) and metalloproteases which are known to play key roles in the pathogenesis of osteoarthritis while exerting no effect on phospholipase A2, cyclooxygenase or lipoxygenase. It showed anti-inflammatory effects on animal models and reduced structural changes in several animal models. Therefore, we investigate the role of diacerein in patients with hand osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Ages over 40 years-old
* Conforming to the classification criteria of American College of Rheumatology*
* More than 1 tender joints
* Self reported hand pain which is more than 30 mm on the Australian/Canadian Osteoarthritis Hand Index visual analogue scales (VAS) after wash out period of 2 weeks

Exclusion Criteria:

* Pregnant or lactating women
* Previous history of hypersensitivity to Diacerein
* Patients who had taken oral corticosteroid or intraarticular steroid to hand joints within 3 months of enrollment
* Patients who were injected with hyaluronic acid to hand joints within 6 months of enrollment
* Patients who underwent surgery in any joints of the hands
* AST/ALT > 2x upper normal range
* Serum Cr > 1.4 mg/dl
* Patients who have severe comorbidities such as severe congestive heart failure or pulmonary disease
* Patients who took oral anticoagulants.
* Patients who refuse to sign the consent form

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Australian/Canadian Osteoarthritis Hand Index (AUSCAN) pain score at 4 week point | 12 weeks

SECONDARY OUTCOMES:
AUSCAN stiffness score at 4 week point | 12wks
AUSCAN pain score at 12 week point | 12wk

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin K, Kim JW, Moon KW, Yang JA, Lee EY, Song YW, Lee EB. The efficacy of diacerein in hand osteoarthritis: a double-blind, randomized, placebo-controlled study. Clin Ther. 2013 Apr;35(4):431-9. doi: 10.1016/j.clinthera.2013.02.009. Epub 2013 Mar 6. PMID 23474153